CLINICAL TRIAL: NCT03293485
Title: A Phase III Non-randomized, Non-controlled, Open Label Clinical Trial to Study the Safety and Efficacy of Imipenem/Cilastatin/Relebactam (IMI/REL [MK-7655A]) in Japanese Subjects With Complicated Intra-Abdominal Infection (cIAI) or Complicated Urinary Tract Infection (cUTI)
Brief Title: Efficacy and Safety of Imipenem+Cilastatin/Relebactam (MK-7655A) in Japanese Participants With Complicated Intra-abdominal Infection or Complicated Urinary Tract Infection (MK-7655A-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7655A-017; 173738 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2017-09-15; First posted 2017-09-26 (Actual); Results first posted 2019-09-17 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Complicated Intra-abdominal Infection; Complicated Urinary Tract Infection
MeSH Terms: interventions — imipenem, cilastatin and relebactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Imipenem+Cilastatin/Relebactam (Experimental): Participants with cIAI or cUTI will receive imipenem+cilastatin/relebactam intravenous (IV) infusion once every 6 hours for 5 to 14 days
  Interventions: Drug: Imipenem+Cilastatin/Relebactam

INTERVENTIONS:
Drug: Imipenem+Cilastatin/Relebactam — Imipenem+Cilastatin/Relebactam 200/100 mg to 500/250 mg, depending on renal function, 30-minute IV infusion once every 6 hours
  Other Names: IMI/REL; MK-7655A

SUMMARY:
The study will evaluate the efficacy and safety of imipenem+cilastatin/relebactam (IMI/REL, MK-7655A) in Japanese participants with complicated intra-abdominal infection (cIAI) or complicated urinary tract infection (cUTI).

ELIGIBILITY:
Inclusion Criteria:

* requires hospitalization and treatment with IV antibiotic therapy for complicated intraabdominal infection (cIAI) or complicated urinary tract infection (cUTI). Per-protocol diagnostic criteria apply to the qualifying infection types.
* infection is known or thought to be caused by microorganisms susceptible to the IV study therapy
* baseline specimen for primary infection site culture obtained at operative procedure in Screening period or at Baseline for cIAI participants, and within 48 hours before initiation of IV study drug for cUTI participants
* female or male who is not of reproductive potential, or female or male who is of reproductive potential and agrees to avoid becoming pregnant or impregnating a partner from the time of consent through completion of the study, by practicing abstinence from heterosexual activity or using acceptable contraception during heterosexual activity.

Exclusion Criteria:

* received any amount of effective antibiotic therapy after obtaining the culture for admission to the study and before administration of the first dose of IV study therapy
* received treatment with systemic effective antibiotics for >24 hours within the 72 hours before initiation of study therapy
* has a concurrent infection, including endocarditis, osteomyelitis, meningitis, or prosthetic joint infection, that would interfere with evaluation of response to IMI/REL
* has a cIAI or cUTI due to a confirmed fungal pathogen
* has a cUTI that meets any of the following: 1) complete obstruction of any portion of the urinary tract, 2) known ileal loop, 3) intractable vesico-ureteral reflux, 4) presence of indwelling urinary catheter which cannot be removed at study entry
* has a cIAI that meets any of the following: 1) infection that should be managed by Staged Abdominal Repair (STAR) or open abdomen therapy, 2) infection limited to the hollow viscus
* history of serious allergy, hypersensitivity, or any serious reaction to any carbapenem, cephalosporin, penicillin or other beta-lactam agent, or other beta-lactamase inhibitors
* female who is pregnant or is expecting to conceive, is breastfeeding, or plans to breastfeed before completion of the study
* history of a seizure disorder
* anticipates to be treated with valproic acid, concomitant IV or an oral antimicrobial considered effective to the index pathogen, in addition to the study treatment
* is receiving immunosuppressive therapy, including high-dose corticosteroids
* is undergoing hemodialysis or peritoneal dialysis
* participated in any other clinical study involving an investigational or experimental medication during the previous 30 days before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- Japan (29):
  - Nagoya Ekisaikai Hospital ( Site 1724), Nagoya, Aichi-ken
  - Toyota Memorial Hospital ( Site 1708), Toyota, Aichi-ken
  - Medical Corporation Chiyukai Fukuoka Shin Mizumaki Hospital ( Site 1710), Onga-gun, Fukuoka
  - Shin Yukuhashi Hospital ( Site 1722), Yukuhashi, Fukuoka
  - National Hospital Organization Fukuyama Medical Center ( Site 1706), Fukuyama, Hiroshima
  - Fukuyama City Hospital ( Site 1721), Fukuyama, Hiroshima
  - KKR Sapporo Medical Center ( Site 1728), Sapporo, Hokkaido
  - Sano Hospital ( Site 1701), Kobe, Hyōgo
  - National Hospital Organization Mito Medical Center ( Site 1729), Higashiibaraki-gun, Ibaraki
  - Medical Corporation Tokushukai Koga General Hospital ( Site 1712), Koga, Ibaraki
  - Ishikawa Prefectural Central Hospital ( Site 1707), Kanazawa, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center ( Site 1716), Kanazawa, Ishikawa-ken
  - Kawahara Clinic ( Site 1719), Aira, Kagoshima-ken
  - National Hospital Organization Yokohama Medical Center ( Site 1702), Yokohama, Kanagawa
  - National Hospital Organization Mie Chuo Medical Center ( Site 1727), Tsu, Mie-ken
  - Japan Labour Health And Safety Organization Tohoku Rosai Hospital ( Site 1714), Sendai, Miyagi
  - National Hospital Organization Sendai Medical Center ( Site 1723), Sendai, Miyagi
  - Suwa Red Cross Hospital ( Site 1705), Suwa, Nagano
  - National Hospital Organization Nagasaki Medical Center ( Site 1718), Ōmura, Nagasaki
  - National Hospital Organization Osaka Minami Medical Center ( Site 1715), Kawachi-Nagano, Osaka
  - National Hospital Organization Utsunomiya National Hospital ( Site 1711), Utsunomiya, Tochigi
  - National Hospital Organization Minami Wakayama Medical Center ( Site 1725), Tanabe, Wakayama
  - Yamanashi Prefectural Central Hospital ( Site 1703), Kofu, Yamanashi
  - Fukuiken Saiseikai Hospital ( Site 1704), Fukui
  - Medical Corporation Chiyukai Fukuoka Wajiro Hospital ( Site 1709), Fukuoka
  - Medical Corporation Shingenkai Kawahara Urological Clinic ( Site 1726), Kagoshima
  - Medical Corporation Seifukai Yagi Clinic ( Site 1720), Kagoshima
  - National Hospital Organization Kumamoto Medical Center ( Site 1713), Kumamoto
  - National Hospital Organization Oita Medical Center ( Site 1717), Ōita

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kohno S, Bando H, Yoneyama F, Kikukawa H, Kawahara K, Shirakawa M, Aoyama N, Brown M, Paschke A, Takase A. The safety and efficacy of relebactam/imipenem/cilastatin in Japanese patients with complicated intra-abdominal infection or complicated urinary tract infection: A multicenter, open-label, noncomparative phase 3 study. J Infect Chemother. 2021 Feb;27(2):262-270. doi: 10.1016/j.jiac.2020.09.032. Epub 2020 Nov 13. PMID 33191112

RESULTS

PARTICIPANT FLOW:
Groups:
- cIAI/cUTI: Participants with complicated intra-abdominal infection (cIAI) or complicated urinary tract infection (cUTI) received intravenous imipenem+cilastatin+relebactam (IMI/REL) once every 6 hours for 5-14 days.
Period: Overall Study
Arm/Group | cIAI/cUTI
Started | 83
Treated | 81
Completed | 78
Not Completed | 5
Not completed — Death | 1
Not completed — Screen Failure | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- cIAI/cUTI: Participants with cIAI or cUTI received intravenous imipenem+cilastatin+relebactam once every 6 hours for 5-14 days.
Arm/Group | cIAI/cUTI
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 83
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Infection Type [Count of Participants; unit: Participants] — Participants enrolled with either complicated intra-abdominal infection (cIAI), or complicated urinary tract infection (cUTI).
  Participants
    cIAI | 39
    cUTI | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AE)
Description: The percentage of participants experiencing ≥1 AE was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to 28 days
Population: Per protocol, the population analyzed was all participants who received ≥1 dose of intravenous imipenem+cilastatin+relebactam.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | cIAI/cUTI
Number analyzed (Participants) | 81
Percentage of Participants | 74.1 [63.5 to 82.4]

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: The percentage of participants who discontinued from study medication due to an adverse event was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to 14 days (End of Therapy Visit)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | cIAI/cUTI
Number analyzed (Participants) | 81
Percentage of Participants | 4.9 [1.6 to 12.4]

3. Primary Outcome: Percentage of Complicated Intra-Abdominal Infection (cIAI) Participants With Favorable Clinical Response at End of Therapy Visit
Description: The percentage of participants with cIAI who display a favorable clinical response at End of Therapy visit was presented. Per protocol, a subset of the cIAI/cUTI study arm was analyzed: only participants with cIAI were evaluated because clinical response is primarily relevant to cIAI. Favorable clinical response is a rating of "cure" or "improved" as determined by the investigator at the End of Therapy Visit. "Cure" is defined as: all pretherapy signs and symptoms of the index infection(s) have resolved (or returned to preinfection status) AND no additional intravenous antibiotic therapy is required AND no unplanned surgical or percutaneous drainage procedures have been performed. "Improved" is defined as: All or most pretherapy signs and symptoms of the index infection(s) have improved or resolved (or returned to preinfection status) AND no additional intravenous antibiotic therapy is required AND no unplanned surgical or percutaneous drainage procedures have been performed.
Time Frame: Between Day 5 and Day 14 (End of Therapy Visit)
Population: Per protocol, the population analyzed was all participants with cIAI who received intravenous imipenem+cilastatin+relebactam ≥96 hours, whose pre-study infection-site culture grew ≥1 gram-negative enteric and/or anaerobic pathogen, and who had no major deviations from the protocol that may substantially affect the results of the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- cIAI: Participants with cIAI received intravenous imipenem+cilastatin+relebactam once every 6 hours for 5-14 days.
Arm/Group | cIAI
Number analyzed (Participants) | 28
Percentage of Participants | 85.7 [67.9 to 94.9]

4. Primary Outcome: Percentage of Complicated Urinary Tract Infection (cUTI) Participants With Favorable Overall Microbiological Response at End of Therapy Visit
Description: The percentage of participants with cUTI who display a favorable Overall Microbiological Response at the End of Therapy visit was calculated. Per protocol, only a subset of the cIAI/cUTI study arm was analyzed: only participants with cUTI were evaluated because the microbiological response evaluation is primarily relevant to cUTI. A favorable Overall Microbiological Response is defined as a urine culture taken at the End of Therapy Visit showing eradication (e.g., ≥10^5 CFU/mL is reduced to <10^4 CFU/mL) of all uropathogens found at study entry.
Time Frame: Between Day 5 and Day 14 (End of Therapy Visit)
Population: Per protocol, the population analyzed was all participants with cUTI who received intravenous imipenem+cilastatin+relebactam ≥96 hours, whose pre-study infection-site culture grew ≥1 gram-negative and/or anaerobic pathogen, and who had no major deviations from the protocol that may substantially affect the results of the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- cUTI: Participants with cUTI received intravenous imipenem+cilastatin+relebactam once every 6 hours for 5-14 days.
Arm/Group | cUTI
Number analyzed (Participants) | 39
Percentage of Participants | 100 [89.3 to 100.0]

5. Secondary Outcome: Percentage of Complicated Intra-Abdominal Infection (cIAI) Participants With Favorable Clinical Response at Test of Cure Visit
Description: The percentage of participants with cIAI who display a favorable Clinical Response at the Test of Cure visit was calculated. Per protocol, only a subset of the cIAI/cUTI study arm was analyzed: only participants with cIAI were evaluated because the clinical response evaluation is primarily relevant to cIAI. A favorable clinical response is a rating of "cure" as determined by the investigator at the Test of Cure Visit. "Cure" is defined as: all pretherapy signs and symptoms of the index infection(s) have resolved (or returned to "preinfection status") AND no additional intravenous antibiotic therapy is required AND no unplanned surgical or percutaneous drainage procedures have been performed.
Time Frame: Between Day 10 and Day 23 (Test of Cure Visit)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | cIAI
Number analyzed (Participants) | 28
Percentage of Participants | 82.1 [63.9 to 92.6]

6. Secondary Outcome: Percentage of Complicated Urinary Tract Infection (cUTI) Participants With Favorable Overall Microbiological Response at Test of Cure Visit
Description: The percentage of participants with cUTI who display a favorable Overall Microbiological Response at the Test of Cure visit was calculated. Per protocol, only a subset of the cIAI/cUTI study arm was analyzed: only participants with cUTI were evaluated because the microbiological response evaluation is primarily relevant to cUTI. A favorable Overall Microbiological Response is defined as a urine culture taken at the Test of Cure visit still showing eradication (e.g., ≥10^5 CFU/mL is reduced to <10^4 CFU/mL) of all uropathogens found at study entry.
Time Frame: Between Day 10 and Day 23 (Test of Cure Visit)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | cUTI
Number analyzed (Participants) | 39
Percentage of Participants | 59.0 [43.4 to 72.9]

ADVERSE EVENTS:
Time Frame: Up to 28 days (up to 14 days after completion of intravenous study therapy)
Description: Adverse events were reported for all participants who received at least one dose of IV study therapy.
Arm/Group | cIAI/cUTI
All-Cause Mortality (participants affected / at risk) | 1/81
Serious Adverse Events (participants affected / at risk) | 9/81
Other Adverse Events (participants affected / at risk) | 18/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cIAI/cUTI (N=81)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2)
Pelvic abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cIAI/cUTI (N=81)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (9)
Nasopharyngitis (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication (or after public disclosure of the results at www.clinicaltrials.gov if multicenter manuscript is not planned), an investigator and colleagues may publish their data independently.

Sponsor must have opportunity to review proposed abstracts, manuscripts or presentations 45 days prior to submission for publication/presentation. Confidential information must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03293485/Prot_SAP_000.pdf